CLINICAL TRIAL: NCT05520892
Title: A Multicenter, Randomized Controlled Study of Two Regimens of Intravenous Immune Globulin in the Treatment of Newly Diagnosed Immune Thrombocytopenia in Children
Brief Title: Two Regimens of IVIG in the Treatment of Newly Diagnosed ITP in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Quanzhou First Hospital (Other); Nanping First Hospital Affiliated to Fujian Medical University (Unknown); The Second Hospital of Anhui Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Longyan City First Hospital (Other); The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022YF024-01
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-02

CONDITIONS: Newly Diagnosed Immune Thrombocytopenia in Children, First Line Treatment
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low-dose intravenous immunoglobulin (Experimental): 0.4g/kg.d, d1-5
  Interventions: Drug: intravenous immunoglobulin
- high-dose intravenous immunoglobulin (Active Comparator): 1.0g/kg.d, d1-2
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Drug: intravenous immunoglobulin — To compare the efficacy of two different dosage regimens of intravenous immune globulin (IVIG) in the treatment of children with newly diagnosed immune thrombocytopenia

SUMMARY:
To compare the efficacy of two different dosage regimens of intravenous immune globulin (IVIG) in the treatment of children with newly diagnosed immune thrombocytopenia, and to reduce related adverse reactions and economic burdens on the premise of ensuring the remission rate

ELIGIBILITY:
Inclusion Criteria:Subjects enrolled in this study must meet all of the following criteria:

1. Meet the diagnostic criteria of ITP and be diagnosed for the first time without treatment
2. Age > 28 days and ≤ 14 years old
3. PLT<20×109/L
4. Have signed the informed consent

Exclusion Criteria:Anyone who has any of the following conditions will not enter the clinical study:

1. Intracranial hemorrhage or severe gastrointestinal or urinary tract hemorrhage requiring emergency treatment, such as simultaneous use of platelet transfusion and glucocorticoid therapy
2. Received glucocorticoid or IVIG therapy within 6 months
3. Weight > 40kg
4. Menstrual female patients
5. Patients with underlying diseases such as tumor diseases, autoimmune diseases or genetic diseases
6. Patients who have received radiotherapy and chemotherapy
7. There are any significant abnormal coexisting diseases or mental illnesses that affect the patient's life safety and compliance, and affect informed consent, research participation, follow-up or interpretation of results -

Ages: 29 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 580 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
early response to treatment | 7 days after treatment
  Platelet counts after 7 days of IVIG treatment

SECONDARY OUTCOMES:
Economic Indicators | 1 week
  Calculate the total amount of IVIG used in 1 week (weight normalized)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 week
  Incidence of Treatment-Emergent Adverse Events in 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Children with newly dignosed ITP, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No